CLINICAL TRIAL: NCT04555564
Title: Tc99m-Macroaggregated Albumin Bronchial Artery Injection During Bronchial Embolization for Pulmonary Mass Induced Hemoptysis for Dosimetry Planning
Brief Title: Tc99m Macroaggregated Albumin Bronchial Artery Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn in IRB
Sponsor: Johns Hopkins University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00222311
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2021-08

CONDITIONS: Hemoptysis; Malignant Neoplasm; Lung Cancer
Keywords: Lung cancer; lung metastasis; Bronchial artery embolization; MAA study; Dosimetry
MeSH Terms: conditions — Hemoptysis; Neoplasms; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm, prospective, single-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Technicium 99 MAA (Experimental): Participants will receive bronchial artery administration of Technicium 99 MAA
  Interventions: Procedure: Technicium 99 MAA infusion

INTERVENTIONS:
Procedure: Technicium 99 MAA infusion — 4mci of Technicium 99 MAA will be infused into the bronchial artery via a catheter prior to a standard therapy (bronchial artery embolization). The patient will undergo nuclear medicine imaging following this intervention to quantify MAA distribution within the lung tumor and adjacent lung tissue.

SUMMARY:
This is a single-arm, single-center, prospective pilot study to perform bronchial artery Tc-99m-MAA infusion to determine the predicted whole lung versus lung tumor dosimetry of a possible intra-arterial radioembolization.

DETAILED DESCRIPTION:
This study is a prospective, single-arm pilot study for patients presenting with hemoptysis from lung cancers. Prior to a therapeutic bronchial artery embolization (standard therapy), Tc99m-MAA will be administered to the bronchial artery and an imaging will be obtained to determine the distribution of MAA.

The primary objective will be quantification of Tc99m-MAA uptake within the tumor and surrounding structures (esophagus, bronchi, pericardium, spine). This is a purely descriptive study and no statistical comparison or correlation will be made. Dosimetry will be reported for each patient, as well as range and mean with standard deviation. Additional activity calculation methods and reporting metrics may additionally be used. Non-statistical comparison will be made to literature-reported external-beam radiation dose-related tumor response and adjacent-organ toxicities to develop a preliminary assessment of the potential for efficacy and anticipated safety-profile of Yittrium-90 bronchial artery radio-embolization.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age and older
* Patients with known active lung cancer with a history of prior hemoptysis presenting for bronchial artery embolization will be considered.
* Patients must be presenting for secondary prophylaxis of hemoptysis
* Willing and able to understand and sign a written informed consent document.
* Willing and able to undergo all study procedures.

Exclusion Criteria:

* Patients with current active hemoptysis
* Any acute or chronic inflammatory disease or medical conditions that in the investigator's opinion may interfere with the study procedures or the interpretation of the study results.
* If female, not of childbearing potential or negative serum β-human chorionic gonadotropin pregnancy test prior to radiotracer injection.
* If female, not nursing.
* Subjects who have exclusion criteria that would prevent them from receiving a CT scan or fluoroscopy, or administration of contrast.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to macro-aggregated albumin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of Tc99m-MAA uptake | 12 months
  The primary objective will be quantification of Tc99m-MAA uptake (measured in "Gray") within the tumor and surrounding structures (esophagus, bronchi, pericardium, spine). This is a purely descriptive study and no statistical comparison or correlation will be made. This assessment will be done for each participant at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Buethe, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chun JY, Belli AM. Immediate and long-term outcomes of bronchial and non-bronchial systemic artery embolisation for the management of haemoptysis. Eur Radiol. 2010 Mar;20(3):558-65. doi: 10.1007/s00330-009-1591-3. Epub 2009 Sep 2. PMID 19727742
- [Background] Wang GR, Ensor JE, Gupta S, Hicks ME, Tam AL. Bronchial artery embolization for the management of hemoptysis in oncology patients: utility and prognostic factors. J Vasc Interv Radiol. 2009 Jun;20(6):722-9. doi: 10.1016/j.jvir.2009.02.016. Epub 2009 May 5. PMID 19406667
- [Background] Swanson KL, Johnson CM, Prakash UB, McKusick MA, Andrews JC, Stanson AW. Bronchial artery embolization : experience with 54 patients. Chest. 2002 Mar;121(3):789-95. doi: 10.1378/chest.121.3.789. PMID 11888961
- [Background] Eldridge L, Moldobaeva A, Zhong Q, Jenkins J, Snyder M, Brown RH, Mitzner W, Wagner EM. Bronchial Artery Angiogenesis Drives Lung Tumor Growth. Cancer Res. 2016 Oct 15;76(20):5962-5969. doi: 10.1158/0008-5472.CAN-16-1131. Epub 2016 Aug 28. PMID 27569207
- [Background] Jonas AM, Carrington CB. Vascular patterns in primary and secondary pulmonary tumors in the dog. Am J Pathol. 1969 Jul;56(1):79-95. No abstract available. PMID 4893319
- [Background] CUDKOWICZ L, ARMSTRONG JB. The blood supply of malignant pulmonary neoplasms. Thorax. 1953 Jun;8(2):153-6. doi: 10.1136/thx.8.2.152. No abstract available. PMID 13077512
- [Background] Ricke J, Grosser O, Amthauer H. Y90-radioembolization of lung metastases via the bronchial artery: a report of 2 cases. Cardiovasc Intervent Radiol. 2013 Dec;36(6):1664-1669. doi: 10.1007/s00270-013-0690-3. Epub 2013 Jul 10. PMID 23839007